CLINICAL TRIAL: NCT05279807
Title: Interventional Clinical Trial to Assess Efficacy and Safety of the Extemporaneous Combination of Zofenopril Calcium and Amlodipine in Grade 1-2 Hypertensive Patients Versus Each Monotherapy - (MASOLINO Study)
Brief Title: Effectiveness and Safety of Combination of Amlodipine and Zofenopril in Hypertensive Patients Versus Each Monotherapy
Acronym: Masolino
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini International Operations Luxembourg SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEIN/20/ZoAm-Hyp/001
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2022-08

CONDITIONS: Hypertension
Keywords: Hypertension; Combination Therapy; Zofenopril; Nebivolol; Fixed Dose Combination
MeSH Terms: conditions — Hypertension | interventions — zofenopril; Amlodipine

STUDY DESIGN:
Intervention Model Description: Patients with uncontrolled BP on treatment with any Ace-i or any CCB, if eligible, will enter a 4-week run-in period.
  Patients will then be all assigned to mono-therapy with ZOF 30mg or AML 5mg for 4 weeks if in treatment with Ace-i or CCB respectively.
  At Visit 2 patients with uncontrolled BP, tolerating treatment and with adherence within 80%/120% ranges, will receive extemporaneous combination ZOF 30mg+AML 5mg, while patients with controlled BP, tolerating treatment or with adherence out of 80%/120% range, will be withdrawn from the study together with patients with SBP/DBP ≥ 180/100 mmHg.
  At Visit 3 (Visit 2 + 4 weeks ± 2 days) controlled patients will continue extemporaneous combination for additional 4 weeks ± 2 days, while uncontrolled patients will be up-titrated to ZOF 30mg/AML 10mg for the same time. Patients with SBP/DBP ≥ 180/100 mmHg or not tolerating extemporaneous combination or with adherence out of 80%/120% range, will be withdrawn from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zofenopril 30 mg (Active Comparator): Single dose Phase (4 weeks): patients will be treated with Zofenopril 30 mg. Combination Phase (8 weeks) uncontrolled patients will be treated with the extemporaneous combination of Zofenopril 30 mg and Amlodipine 5mg for 4 weeks. Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks while controlled patients with Zofenopril 30mg/Amlodipine 5mg will continue with the same therapy.
  Interventions: Drug: Zofenopril; Drug: Amlodipine
- Amlodipine 5/10 mg (Active Comparator): Single dose Phase (4 weeks): patients will be treated with Amlodipine 5 mg. Combination Phase (8 weeks) uncontrolled patients will be treated with the extemporaneous combination of Zofenopril 30 mg and Amlodipine 5mg for 4 weeks. Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks while controlled patients with Zofenopril 30mg/Amlodipine 5mg will continue with the same therapy.
  Interventions: Drug: Zofenopril; Drug: Amlodipine

INTERVENTIONS:
Drug: Zofenopril — Film-Coated tablets administered orally once daily according instructions provided by Principal Investigator.
Drug: Amlodipine — Tablets of 5mg and 10mg administered orally once daily according instructions provided by Principal Investigator.

SUMMARY:
Study to assess the anti-hypertensive efficacy and safety of the extemporaneous combination of Zofenopril 30 mg in combination with Amlodipine 5 mg or AML 10 mg in lowering the sitting diastolic BP after 8 weeks of treatment in patients with uncontrolled BP previously treated with Zofenopril or Amlodipine (5 mg) monotherapies for at least 4 weeks.

DETAILED DESCRIPTION:
Approximately 290 patients are planned to be screened to ensure at least 216 patients complete the run-in period and start with the assessment period.

Patients with Grade 1-2 hypertensive patients (blood pressure [BP] ranging from ≥140/90 mmHg to ≤179/109 mmHg) on treatment with any angiotensin converting enzyme inhibitors (ACE-i) including Zofenopril (ZOF)30 mg or with calcium channel blockers (CCBs) including Amlodipine (AML)5 mg will be screened for eligibility (Visit 1).

Allowed CCBs: Felodipine, isradipine, lacidipine, lercanidipine, nicardipine, nifedipine, and nisoldipine. Patients treated with other dosages of ZOF (other than 30 mg) are not allowed to be screened. After screening, on the same day, eligible patients, will enter into a 4-week run-in period, during which patients on other ACE-i will be assigned to monotherapy with ZOF 30 mg while patients on CCBs will be assigned to monotherapy with AML 5 mg for 4 weeks. Patients with on-going treatment zofenopril 30 mg and amlodipine 5mg will continue on the same treatment for 4 weeks.

After the run-in period (4 weeks ± 2 days), BP will be further assessed (Visit 2), if BP levels are over the defined controlled target goal, sitting Systolic Blood Pressure (SBP)/Diastolic Blood Pressure (DBP) >130/80 mmHg, treatment is well tolerated and adherence to the treatments ranges from 80% to 120%, patients will enter the assessment period, where they will be assigned to the extemporaneous combination of ZOF 30 mg and AML 5 mg. At Visit 2 patients with SBP/DBP values classified as Grade 3 (SBP ≥ 180 or DBP ≥ 110 mmHg) hypertension will be withdrawn from the study.

If patients, at Visit 2, after the run-in period, have a controlled BP (sitting SBP/DBP≤130/80 mmHg) or do not tolerate the treatment or have an adherence range below 80% or superior to 120%, they will be withdrawn from the study.

The patients will be assessed for further 8 weeks (assessment period). After 4 weeks ± 2 days from Visit 2,during the assessment period patients receiving the extemporaneous combination of ZOF 30 mg and AML 5 mg, will be further evaluated (Visit 3): controlled patients (sitting SBP/DBP ≤130/80 mmHg) will continue the same extemporaneous combination for additional 4 weeks ± 2 days, while uncontrolled patients (sitting SBP/DBP >130/80 mmHg) will be up-titrated from ZOF/AML 30/5 mg to ZOF/AML 30/10 mg for further 4 weeks ± 2 days. At Visit 3 patients with SBP/DBP values classified as Grade 3 (SBP ≥ 180 or DBP ≥ 110 mmHg) hypertension will be withdrawn from the study. If patients at Visit 3, do not tolerate the extemporaneous combination treatment or they have an adherence range below 80% or superior to 120%, they will be withdrawn from the study.

At the end of the assessment period (8 weeks ± 4 days) at Visit 4, the anti-hypertensive effect of the extemporaneous combination (ZOF/AML 30/5 mg and ZOF/AML 30/10 mg) will be evaluated.

Efforts will be made to achieve 1:1 ratio in the enrolment of patients receiving any ACE-i or allowed CCBs (refer to section Subject Study Phases Duration for allowed CCBs). At Visit 2, a minimum of 45% of uncontrolled patients receiving treatment with ZOF 30 mg or AML 5 mg are required to enter the assessment period, in order to maintain a balance between the 2 treatments during the assessment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Grade 1-2 hypertensive patients: with mean sitting SBP ≥140 mmHg and ≤179 mmHg and/or mean sitting DBP ≥ 90 mmHg and ≤109 mmHg at Screening, with ≥18 and ≤65 years of age, on monotherapy either with ZOF 30 mg or AML 5mg or any other ACE-I or CCBs (Felodipine, isradipine, lacidipine, lercanidipine, nicardipine, nifedipine, and nisoldipine) for at least 1 month before Visit 1 (Screening).
2. Patients who are able to understand and give written informed consent at Screening
3. Patients who are available for the entire trial period and willing to adhere to the protocol requirements
4. Ability to take oral medication and willing to adhere to the drug regimen
5. Female patients are eligible to participate if not pregnant, or not breastfeeding and must refrain from donating or storing eggs. For females of reproductive potential: use of highly effective contraception (e.g., method of birth control throughout the study period and for 4 weeks after study completion defined as a method which results in a failure rate of less than 1% per year) such as:

   * Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
   * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion
   * Vasectomized partner (performed at least 2 months before screening) (if the partner is the sole sexual partner of the trial participant and that the vasectomized partner has received medical assessment of the surgical success)
6. A male patient must agree to use contraception during the whole study period and for at least 1 week after the last dose of study treatment and refrain from donating sperms during this period

Exclusion Criteria:

1. Known contraindications, presence of not recommended/contraindicated concomitant therapy allergies, or significant history of hypersensitivity to zofenopril, amlodipine, other ACE-inhibitors or dihydropyridines, or any related products including excipients of the formulations as outlined in the Investigator's Brochure (IB), or summary of product characteristics (SmPCs) or local package inserts for AML and ZOF
2. Patients with serious disorders (in the opinion of the Investigator) which may limit the ability to evaluate the efficacy or safety of the tested medications, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine/ or metabolic, haematological, or oncological, neurological, and psychiatric diseases. The same applies for immunocompromised and/or neutropenic patients
3. Patients having a history of the following within the last 6 months: myocardial infarction, unstable angina pectoris, percutaneous coronary intervention, bypass surgery, valve replacement (transcatheter aortic valve implantation, mitral-clip),cerebrovascular accident (stroke, heart failure, hypertensive encephalopathy, cerebrovascular accident (stroke), or transient ischemic attack. Patients with who have undergone other surgery that in the in the opinion of the Investigator may limit the ability to evaluate the efficacy or safety of the tested medications.
4. Patients with secondary hypertension of any aetiology such as renal diseases, pheochromocytoma, Cushing's syndrome hyperaldosteronism, renovascular disease, thyroid disorders
5. Patients with severe heart failure (New York Heart Association classification III-IV), a narrowing of the aortic or bicuspid valve, an obstruction of cardiac outflow (obstructive, hypertrophic cardiomyopathy) or symptomatic coronary disease
6. Patients with clinical evidence of renal disease as per the Investigator's judgement (including renovascular occlusive disease, nephrectomy and/or renal transplant, bilateral renal artery stenosis or unilateral renal artery stenosis in a solitary kidney, or severe renal impairment)
7. Patients with history of angioneurotic oedema
8. Patients with clinically relevant hepatic impairment
9. Patients with sick sinus syndrome, including sino-atrial block
10. Patients with second- or third-degree heart block (without a pacemaker)
11. Participation in any other interventional drug trial or exposure to other investigational agents within 30 days before Screening (Visit 1)
12. Inability to cooperate or any condition that, in the opinion of the Investigator, could increase the patient's risk of participating in the study or confound the outcome of the study
13. Patients with conditions that, in the opinion of the Investigator, would prevent a careful adherence to the protocol
14. Patients with severe hypotension
15. Patients who suffer from shock (including cardiogenic shock)
16. Patients treated with Amlodipine 10 mg and Zofenopril (other than 30 mg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Volpe, Professor, Principal Investigator — University "Sapienza" Rome
Locations (1):
- Investigational site, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After Screening visit, eligible patients entered a 4 week run-in period (from week -4 to week 0) on the same day of the screening visit. Patients previously receiving ZOF 30 mg or AML 5 mg continued the same treatment, patients receiving any other angiotensin converting enzyme inhibitors, were switched to ZOF 30 mg, while patients receiving calcium channel blockers received AML 5 mg.
  Assessment period starts from week 0 (baseline) till week 8 for a total of 8 weeks
Groups:
- Zofenopril 30mg: MONOTHERAPY PERIOD (4 weeks): patients will be treated with Zofenopril 30 mg during the Run In period (week -4 to week 0) COMBINATION THERAPY PERIOD: During the Assessment period of 8 weeks (week 0 - week 8) uncontrolled patients will be treated with the extemporaneous combination of Zofenopril 30 mg and Amlodipine 5mg for 4 weeks. Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks while controlled patients with Zofenopril 30mg/Amlodipine 5mg will continue with the same therapy during the Assessment Period (week 0 - week 4).
  Zofenopril: Film-Coated tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 5mg and 10mg administered orally once daily according instructions provided by Principal Investigator.
- Amlodipine 5/10 mg: MONOTHERAPY PERIOD (4 weeks): patients will be treated with Amlodipine 5 mg during the Run In period (week -4 to week 0) COMBINATION THERAPY PERIOD: During the Assessment period of 8 weeks (week 0 - week 8) uncontrolled patients will be treated with the extemporaneous combination of Zofenopril 30 mg and Amlodipine 5mg for 4 weeks. Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks while controlled patients with Zofenopril 30mg/Amlodipine 5mg will continue with the same therapy.
  Zofenopril: Film-Coated tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 5mg and 10mg administered orally once daily according instructions provided by Principal Investigator.
Period: Overall Study
Arm/Group | Zofenopril 30mg | Amlodipine 5/10 mg
Started | 144 | 133
Completed | 142 | 132
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Laboratory Abnormal Results | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Zofenopril 30mg: MONOTHERAPY PERIOD (4 weeks): patients will be treated with Zofenopril30 mg during the Run In period (week -4 to week 0) COMBINATION THERAPY PERIOD: During the Assessment period of 8 weeks (week 0 - week 8) uncontrolled patients will be treated with the extemporaneous combination of Zofenopril 30 mg and Amlodipine 5mg for 4 weeks. Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks while controlled patients with Zofenopril 30mg/Amlodipine 5mg will continue with the same therapy.
  Zofenopril: Film-Coated tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 5mg and 10mg administered orally once daily according instructions provided by Principal Investigator.
- Amlodipine 5/10 mg: MONOTHERAPY PERIOD (4 weeks): patients will be treated with Amlodipine 5 mg. COMBINATION THERAPY PERIOD: During the Assessment period of 8 weeks (week0 - week 8) uncontrolled patients will be treated with the extemporaneous combination of Zofenopril 30 mg and Amlodipine 5mg for 4 weeks. Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks while controlled patients with Zofenopril 30mg/Amlodipine 5mg will continue with the same therapy.
  Zofenopril: Film-Coated tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 5mg and 10mg administered orally once daily according instructions provided by Principal Investigator.
- Total: Total of all reporting groups
Arm/Group | Zofenopril 30mg | Amlodipine 5/10 mg | Total
Number analyzed (Participants) | 144 | 133 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (9.96) | 54.1 (9.03) | 52.3 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 83 | 160
  Male | 67 | 50 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 144 | 133 | 277
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (DBP) Between Visit 2 (Week 0) and Visit 4 (Week 8)
Description: To assess the antihypertensive efficacy of the extemporaneous combination of Zofenopril (ZOF) 30 mg in combination with Amlodipine (AML) 5 mg or AML 10 mg in lowering the sitting diastolic BP between Visit 2 (Week 0) and Visit 4 (Week 8) in patients with uncontrolled BP previously treated with Zofenopril or Amlodipine (5 mg) monotherapies for at least 4 weeks during run-in period.
Time Frame: From Visit 2 (week 0) to Visit 4 (week 8) for a total of 8 weeks
Population: Efficacy Population: all study participants who signed inform consent, met all screening criteria, were enrolled and received at least one dose of the assigned treatment during the run-in period and completed the 4-week run-in period, who met criteria at Visit 2 (Week 0) [uncontrolled BP (sitting Systolic BP/DBP > 130 / 80 mmHg)], tolerated treatment, had treatment adherence between 80 - 120 % and had at least one available post baseline primary efficacy assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Combination Therapy Phase Zofenopril 30mg/Amlodipine 5 or 10 mg: Combination Therapy Phase (8 weeks) from Visit 2 (week 0) to Visit 4 (week 8): uncontrolled patients with Monotherapy (Zofenopril 30mg or Amlodipine 5 mg) are treated with the extemporaneous combination of Zofenopril 30mg and Amlodipine 5mg for 4 weeks. Amlodipine10mg will replace Amlodipine 5mg in uncontrolled patients for further 4 weeks while controlled patients with Zofenopril 30mg/Amlodipine 5mg will continue with the same therapy.
  Zofenopril: Film-Coated tablets administered orally once daily according instructions provided by Principal Investigator.
  Amlodipine: Tablets of 5mg and 10mg administered orally once daily according instructions provided by Principal Investigator.
Arm/Group | Combination Therapy Phase Zofenopril 30mg/Amlodipine 5 or 10 mg
Number analyzed (Participants) | 269
mmHg | -13.5 (8.31)
Statistical Analysis 1: Comparison: Combination Therapy Phase Zofenopril 30mg/Amlodipine 5 or 10 mg; Primary endpoint, verified on the single cohort of patients who completed the monotherapy run-in period, is calculated as the mean difference in sitting diastolic blood pressure between Visit 2 (Week 0, Baseline Visit of the combination therapy) and Visit 4 (Week 8, End of Study Visit). This is not a comparison of two different arms, but a comparison of two measurements taken from the same patient treated with combination therapy (single arm paired pre- vs. post-combination therapy comparison); Test type: Superiority; p < 0.001, Paired Samples T-Test; Mean difference pre vs post treatment = -13.5, 95% CI 2-sided [-14.5 to -12.5]

ADVERSE EVENTS:
Time Frame: From Informed Consent signature at screening visit (Visit 1) occurring 4 week previous than Baseline assessment (Week 0 - Visit 2) to last visit at Week 8 (Visit 4) for an average of 12 weeks. Furthermore patients having any ongoing Adverse Event/Serious Adverse Event at the end of the treatment (Week 8 - Visit 4), will be followed for further 2 weeks via a phone call to check about the status of the Adverse Events/Serious Adverse Events, extending the time frame to a total of 14 weeks.
Description: Safety Population (used for safety analyses): "All study participants enrolled that received at least one dose of the assigned treatment during the run-in period". One Enrolled patient was not dosed and therefore was not part of Safety Population.
  If a patient reports the same Adverse Event (AE) more than once within that System Organ Class/Preferred Term, then that patient will be counted only once for that System Organ Class or Preferred Term
Groups:
- Zofenopril 30mg MONOTHERAPY PERIOD: Patients will be treated with Zofenopril 30 mg during the Run in Period (week -4 to week 0).
  Zofenopril: Film-Coated tablets administered orally once daily according instructions provided by Principal Investigator.
- Amlodipine 5 mg MONOTHERAPY PERIOD: Patients will be treated with Amlodipine 5 mg during the Run in Period (week -4 to week 0).
  Zofenopril: Film-Coated tablets administered orally once daily according instructions provided by Principal Investigator.
- Zofenopril 30mg/Amlodipine 5mg COMBINATION THERAPY PERIOD: Uncontrolled patients at week 0 will be treated with the extemporaneous combination of Zofenopril 30 mg and Amlodipine 5mg for 4 weeks during the Assessment Period (week 0 - week 4).
  Amlodipine: Tablets of 5mg administered orally once daily according instructions provided by Principal Investigator.
- Zofenopril 30mg/Amlodipine 10mg COMBINATION THERAPY PERIOD: Amlodipine 10mg will replace Amlodipine 5mg in uncontrolled patients at week 4 (Visit 3) during the Assessment Period for further 4 weeks (week 4 - week 8) while controlled patients with Zofenopril 30mg/Amlodipine 5mg will continue with the same therapy.
  Amlodipine: Tablets of 10mg administered orally once daily according instructions provided by Principal Investigator.
Arm/Group | Zofenopril 30mg MONOTHERAPY PERIOD | Amlodipine 5 mg MONOTHERAPY PERIOD | Zofenopril 30mg/Amlodipine 5mg COMBINATION THERAPY PERIOD | Zofenopril 30mg/Amlodipine 10mg COMBINATION THERAPY PERIOD
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/133 | 0/149 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/133 | 0/149 | 1/122
Other Adverse Events (participants affected / at risk) | 8/143 | 11/133 | 10/149 | 20/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zofenopril 30mg MONOTHERAPY PERIOD (N=143) | Amlodipine 5 mg MONOTHERAPY PERIOD (N=133) | Zofenopril 30mg/Amlodipine 5mg COMBINATION THERAPY PERIOD (N=149) | Zofenopril 30mg/Amlodipine 10mg COMBINATION THERAPY PERIOD (N=122)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zofenopril 30mg MONOTHERAPY PERIOD (N=143) | Amlodipine 5 mg MONOTHERAPY PERIOD (N=133) | Zofenopril 30mg/Amlodipine 5mg COMBINATION THERAPY PERIOD (N=149) | Zofenopril 30mg/Amlodipine 10mg COMBINATION THERAPY PERIOD (N=122)
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Asthenia (General disorders) | 1 | 2 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 4 | 0 | 4
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 1 | 4
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 6 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT05279807/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT05279807/SAP_001.pdf